CLINICAL TRIAL: NCT05051514
Title: Examination of Postural Stability, Quality of Life, Depression in Patients With Obstructive Sleep Apnea Syndrome
Brief Title: Physical Status of OSA Patients
Acronym: OSASRehab
Status: Completed | Type: Observational
Sponsor: Okan University (Other)
Collaborators: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Tülay Çevik, PT, Assistant Professor, Bitlis Eren University
Other Study IDs: BEU_1
Record Dates: First submitted 2021-04-18; First posted 2021-09-21 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No-Mild Severity OSAS: Mild sleep apnea: An Apnea-Hypopnea Index (AHI) of five to 14 events per hour.
  Interventions: Diagnostic Test: Evaluation
- Moderate to Severe OSAS: Moderate sleep apnea: An Apnea-Hypopnea Index (AHI) of 15 to 29 events per hour.Severe sleep apnea: An Apnea-Hypopnea Index (AHI) of 30 or more events per hour.
  Interventions: Diagnostic Test: Evaluation

INTERVENTIONS:
Diagnostic Test: Evaluation — To examine the differences in postural stability, anxiety/depression, and quality of life of the patients according to the severity of Obstructive Sleep Apnea Syndrome.

SUMMARY:
To investigate the differences in postural stability, anxiety/depression, and quality of life of the patients according to the severity of Obstructive Sleep Apnea Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Getting a diagnosis of OSAS with polysomnography.
* Agree to participate in the study.

Exclusion Criteria:

* Having respiratory system disease (COPD, asthma, bronchiectasis, lung cancer, etc.).
* Sedative, hypnotic drug intake. Use of medical supplements such as diazepam.
* Hypothyroidism, acromegaly.
* Diagnosis of a psychiatric illness.
* Uncontrolled arrhythmia causing symptoms or hemodynamic impairment.
* Pulmonary edema. Pregnancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary care clinic in Bitlis.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2021-04-18 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Postural stability | Day 1.
  The 30 Seconds Sit to Stand Test is a method used to measure the lower extremity muscle strength and postural stability.

SECONDARY OUTCOMES:
Anxiety and depression | Day 1.
  The Hospital Anxiety and Depression Scale (HADS) is a self-report scale developed to determine the risk levels of patients in terms of anxiety and depression. HADS consists of two subscales, one measuring anxiety, with seven items, and another measuring depression, with seven items, which score separately. Those with a score of 10 and above for the anxiety subscale and those with a score of 7 and above for the depression subscale are defined as high-risk patients.

OTHER OUTCOMES:
Quality of life evaluation | Day 1.
  The Short-form 36 questionaire is used to measure Quality of life assessment of Patients. The 36-Item Short Form (SF-36) is an often used, well-researched, self-reported measure of health. It comprises 36 questions that cover eight domains of health. These; physical function (10 items), social function (2 items), role difficulty due to physical problems (4 items) and emotional problems (3 items), mental health (5 items), vitality (4 items), bodily pain (2 item), general health (5 items).

CONTACTS AND LOCATIONS:
Locations (1):
- Bitlis State Hospital, Bitlis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No